CLINICAL TRIAL: NCT06113133
Title: Assessment of Maximal Oxygen Uptake in Persons Enrolled in Exercise-based Cardiac Rehabilitation
Brief Title: Assessment of Maximal Oxygen Uptake in Cardiac Rehabilitation
Status: Completed | Type: Observational
Sponsor: VIA University College (Other)
Responsible Party: Sponsor
Other Study IDs: 9000035
Record Dates: First submitted 2023-06-22; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Oxygen Consumption
Keywords: Physical fitness; heart disease; oxygen consumption
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maximal oxygen uptake: Measurement of maximal oxygen uptake using < 50-millilitre and 100 millilitre oxygen as a cut-off
  Interventions: Diagnostic Test: measurement of oxygen uptake

INTERVENTIONS:
Diagnostic Test: measurement of oxygen uptake — oxygen uptake is obtained during a maximal exercise test

SUMMARY:
To advance the methodology for evaluating persons with heart disease and their maximal oxygen uptake, the primary aim of this study is to investigate the occurrence of a plateau in oxygen uptake. This plateau will be examined for the purpose of assessing VO2 max in persons enrolled in exercise-based cardiac rehabilitation. Furthermore, this study aims to investigate the age-related respiratory exchange ratio, and rating of perceived exertion, and describe their association with the presence of a plateau.

Heart disease and characteristics for all participants are obtained. Participants underwent a maximal exercise test on an ergometer cycle with direct measurement of oxygen uptake to assess oxygen plateau attainment. This included measurement of the maximal oxygen uptake, respiratory exchange ratio, heart rate and the ratio of perceived exertion (BORG6-20).

DETAILED DESCRIPTION:
Oxygen uptake is measured breath-by-breath by a cardiopulmonary exercise test (CPET), and oxygen and carbon dioxide sensors were calibrated before each test along with the flow sensor, there was calibrated with a 3-litre syringe.

To examine the primary aim, the incidence of a plateau in oxygen uptake was examined by comparing the moving average of the last 15 consecutive breaths with the penultimate 15 breaths and cut-offs at <50 ml and <100 ml of oxygen.

Secondary criteria; Respiratory exchange ratio (RER max), Rating of perceived exertion (BORG RPE max) and heart rate (HR max) are examined to determine if the participant performs the exercise test with a maximal effort to exertion. The respiratory exchange ratio (VCO2/VO2) using age-depending RER cut-offs; 1.10 for ages 40-59 years, 1.06 for ages 60-69 years and +70 years to determine if a maximal effort is provided. There are no recommendations for RER cut-off when participants are aged above 69 years. Therefore, they must reach the RER cut-off 1.06 to be evaluated as maximal effort.

The rating of perceived exertion using the BORG RPE 6-20 scale evaluation > 17 is considered maximal effort. The test was supervised by experienced physiotherapists, an in-house nurse supported if necessary, and a physician was available upon request. Participants and physiotherapists were blinded for VO2 max results from CPET. CPET gas exchange system was operated by an experienced researcher.

Maximal heart rate is rated as a maximal effort by cut-offs calculated as 208 - (0.7 x age in years) according to age group. Using respectively, > 92% and > 89% of the calculated HR max for the age group 40-59 years and the age groups 60-69 years and +70 years to consider maximal effort.

ELIGIBILITY:
Inclusion Criteria:

* participants with heart disease referred to exercise-based cardiac rehabilitation in primary healthcare settings were included

Exclusion Criteria:

* heart-related symptoms according to clinical guidelines that prevent participants from performing a maximal exercise test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are adults with heart diseases such as ischemia, heart failure and after heart valve surgery
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake | Pretest is conducted at the first day in rehabilitation. Posttest is conducted when a participant finish rehabilitation or maximal 1 week after the end of the rehabilitation after 12-weeks
  Cardiopulmonary exercise test by Metalyzer 3B to determine maximal oxygen uptake measured in millimetre oxygen

SECONDARY OUTCOMES:
Respiratory exchange ratio | Respiratory exchange ratio is measured during CPET at pretest the first day in rehabilitation. Posttest is conducted the last week of rehabilitation or maximal 1 week after ending the 12-week program.
  Respiratory exchange ratio is according to the production of carbon dioxide divided by oxygen uptake and is expressed numerically for example 1,05. The highest RER value in the last 1 minute of the test is considered the result
Ratio of perceived exertion | The participants rate their perceived exertion immediately after CPET is finished at pretest the first day in rehabilitation. Posttest is conducted the last week of rehabilitation or maximal 1 week after ending the 12-week program.
  Ratio of perceived exertion is assessed using the BORG scale 6-20, where 20 is the highest score
Maximal heart rate | Heart rate is measured during CPET at pretest the first day in rehabilitation. Posttest is conducted the last week of rehabilitation or maximal 1 week after ending the 12-week program.
  Measurement of the heart rate expressed by beats per minute. The highest HR within the last 1 minute of the test is considered the result.

CONTACTS AND LOCATIONS:
Overall Officials: Maribo, Professor, Study Chair — University of Aarhus
Locations (1):
- Claus Sevel, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No